CLINICAL TRIAL: NCT05727852
Title: Exhaled Breath Proton Mass Spectrometry and Assessment of Endothelial Dysfunction in Patients With Respiratory Diseases
Brief Title: Breath Analysis and Arterial Stiffness in Patients With Respiratory Diseases
Status: Enrolling by invitation | Type: Observational
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: RD-comPV- EMP
Record Dates: First submitted 2023-02-06; First posted 2023-02-14 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-03

CONDITIONS: Chronic Respiratory Diseases; Cystic Fibrosis; Lymphangioleiomyomatosis; Hypersensitivity Pneumonitis; Interstitial Lung Diseases; COPD; Bronchial Asthma
Keywords: Proton-transfer reaction mass spectrometry (PTR-TOF-MS); Exhaled volatile organic compounds (eVOCs); Endothelial function; Arterial stiffness; Cardiovascular disorders; Ventilation disorders; Gas exchange disorders
MeSH Terms: conditions — Cystic Fibrosis; Lymphangioleiomyomatosis; Alveolitis, Extrinsic Allergic; Lung Diseases, Interstitial; Pulmonary Disease, Chronic Obstructive; Asthma; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental: patients with chronic respiratory diseases: Included patients, aged ≥ 18 years, with chronic respiratory diseases: COPD, bronchial asthma, cystic fibrosis, lymphangioleiomyomatosis, hypersensitivity pneumonitis and other interstitial lung diseases.
  Intervention: breath analysis using the Compact PTR-MS proton mass spectrometer by Ionicon (Austria); electrocardiogram (ECG) in one lead with an assessment of the pulse wave using a portable cardiac monitor "CardioQvark"; assessment of arterial stiffness using the VaSera VS-1500N Fukuda Denshi device by non-invasive measurement of blood pressure in four limbs with simultaneous recording of electrocardiogram (ECG), phonocardiogram (PCG) and pulse waves on the carotid, femoral arteries, as well as on the arteries of four limbs.
  Interventions:
  Diagnostic Test: Breath analysis using the Compact PTR-MS proton mass spectrometer; Diagnostic Test: Portable cardiac monitor "CardioQvark"; Diagnostic Test: Assessment of arterial stiffness using the VaSera VS-1500N.
  Interventions: Diagnostic Test: Breath test using the Compact PTR-TOF-MS; Diagnostic Test: Portable cardiac monitor "CardioQvark"; Diagnostic Test: Assessment of arterial stiffness using the VaSera VS-1500N
- Active Comparator: Control: Included subjects, aged ≥ 18 years.
  Intervention: breath analysis using the Compact PTR-MS proton mass spectrometer by Ionicon (Austria); electrocardiogram (ECG) in one lead with an assessment of the pulse wave using a portable cardiac monitor "CardioQvark"; assessment of arterial stiffness using the VaSera VS-1500N Fukuda Denshi device by non-invasive measurement of blood pressure in four limbs with simultaneous recording of ECG, phonocardiogram (PCG) and pulse waves on the carotid, femoral arteries, as well as on the arteries of four limbs.
  Interventions:
  Diagnostic Test: Breath analysis using the Compact PTR-MS proton mass spectrometer; Diagnostic Test: Portable cardiac monitor "CardioQvark"; Diagnostic Test: Assessment of arterial stiffness using the VaSera VS-1500N.
  Interventions: Diagnostic Test: Breath test using the Compact PTR-TOF-MS; Diagnostic Test: Portable cardiac monitor "CardioQvark"; Diagnostic Test: Assessment of arterial stiffness using the VaSera VS-1500N

INTERVENTIONS:
Diagnostic Test: Breath test using the Compact PTR-TOF-MS — Breath samples will be analyzed with a proton-transfer reaction mass spectrometer (Compact PTR-MS, Ionicon, Austria) to obtain eVOCs profiles listed as ions at various mass-to-charge ratios (m/z).
Diagnostic Test: Portable cardiac monitor "CardioQvark" — Record an electrocardiogram (ECG) in one lead with an assessment of the pulse wave using a portable cardiac monitor "CardioQvark" (Russia, LLC "L Card" , RU No. RZN 2019/8124 dated February 15, 2019) once. Devices automatically transfer data to the A&D Connect app paired with it (link). When transferring data, they are completely protected. The data obtained using the application must be sent to the specialists of the research group in a depersonalized form.
Diagnostic Test: Assessment of arterial stiffness using the VaSera VS-1500N — Assessment of arterial stiffness using the VaSera VS-1500N Fukuda Denshi device by non-invasive measurement of blood pressure in four limbs with simultaneous recording of ECG, PCG and pulse waves on the carotid, femoral arteries, as well as on the arteries of four limbs.

SUMMARY:
Assessment of cardiovascular disorders using echocardiography and arterial stiffness; comparative noninvasive assessment of volatile organic compound (eVOC) exhale breath patterns in patients with different chronic respiratory diseases with age and gender-matched healthy adults in order to identify a disease-specific exhaled eVOCs profiles and markers of respiratory and cardiovascular disorders.

DETAILED DESCRIPTION:
Evaluating of eVOCs profiles by proton mass spectrometry with a time-of-flight (PTR-TOF) in patients with different chronic respiratory diseases is of great interest for assessing the prognosis and development of severe ventilation and cardiovascular disorders.

The aim of our study is to determine the diagnostic significance of PTR-TOF analysis in patients with chronic respiratory diseases and to identify specific eVOC markers of a severe ventilation and cardiovascular disorders in patients with different chronic respiratory diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent to participate in the study;
2. Age 18 and over;
3. Clinical diagnosis of one of chronic respiratory diseases (COPD, bronchial asthma, cystic fibrosis, lymphangioleiomyomatosis, hypersensitivity pneumonitis or other interstitial lung disease).

Exclusion Criteria:

1. Unable to sign informed consent;
2. Respiratory disease (for controls);
3. Mental illness (severe dementia, schizophrenia, severe depression, manic-depressive psychosis);
4. Acute coronary syndrome, acute cerebrovascular accident, pulmonary embolism within the last 3 months;
5. Oncology;
6. Previous lung transplantation (for patients with respiratory diseases);
7. Diseases and conditions that can change the ECG picture and complicate the analysis of the ECG (conduction disturbance, pacemaker);
8. Inability to use a heart monitor (congenital developmental anomalies, traumatic amputation of the upper limbs, essential tremor, Parkinson's disease);
9. Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of all males and females over 18 years old in the community according to inclusion, non-inclusion, and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-01-30 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Molecular composition of exhaled breath analysed by proton-transfer reaction mass spectrometer (Compact PTR-MS, Ionicon, Austria) | up to 3 years
  Exhaled volatile organic compounds (eVOCs) profiles listed as ions at various mass-to-charge ratios (m/z)
Results of recording an electrocardiogram (ECG) in one lead with an assessment of the pulse wave | up to 3 years
  Pulse wave velocity, augmentation index, pulse wave type (A, B or C) analysed by a portable cardiac monitor "CardioQvark"
Indicators of arterial stiffness | up to 3 years
  Cardio-ankle vascular index and ankle-brachial index analysed with using the VaSera VS-1500N

SECONDARY OUTCOMES:
Composite of clinical records | up to 3 years
  Clinical data are assessed via questionaire according to the Modified Medical Research Council (mMRC) Dyspnea Scale (scale points: 0 scores - the best outcome, 4 scores - the worst outcome) and Borg Dyspnea scale (scale points: 1 score - the best outcome, 10 scores - thr worst outcome), Standard examination of respiratory function (spirometry: FVC, FEV1, FEV1/FVC, FEF75 - % of predicted, absolute value, z-score; body plethysmography: TLC, RV, VC - % of predicted, absolute value, z-score; diffusion test: DLCO, DLCO/VA - % of predicted, absolute value, z-score), echocardiography, CT scan of the chest, if necessary, sputum culture results

CONTACTS AND LOCATIONS:
Locations (1):
- I.M. Sechenov First Moscow State Medical University (Sechenov University), Center "Digital biodesign and personalized healthcare", Moscow, Russia